CLINICAL TRIAL: NCT00796419
Title: Phase III Study Comparing Albumin and Hetastarch Therapy in Acute Lung Injury
Brief Title: Comparative Evaluation of Albumin and Starch Effects in Acute Lung Injury (ALI)
Acronym: CEASE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Greg S. Martin, M.D., M.Sc., Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00002187; R01FD003440 (FDA); 622-2000 (Other: Emory University)
Record Dates: First submitted 2008-11-21; First posted 2008-11-24 (Estimated); Results first posted 2017-04-28 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-03

CONDITIONS: Lung Injury, Acute (ALI); Respiratory Distress Syndrome, Acute (ARDS)
Keywords: Acute lung injury (ALI); Acute respiratory distress syndrome (ARDS); Respiratory failure
MeSH Terms: conditions — Lung Injury; Respiratory Distress Syndrome; Acute Lung Injury; Respiratory Insufficiency | interventions — Serum Albumin, Human; Hydroxyethyl Starch Derivatives

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Intravenous 5% human albumin
  Interventions: Drug: 5% human albumin
- 2 (Experimental): Intravenous 6% hetastarch
  Interventions: Drug: 6% hetastarch

INTERVENTIONS:
Drug: 5% human albumin — Intravenous administration of 250 milliliters (mL) 5% human albumin every 8 hours for 5 days
  Arms: 1
Drug: 6% hetastarch — Intravenous administration of 250mL 6% hetastarch every 8 hours for 5 days
  Arms: 2

SUMMARY:
Acute lung injury (ALI) and acute respiratory distress syndrome (ARDS) are similar conditions in which the lungs are critically injured by another inflammatory process in the body. Together they affect more than 150,000 people per year in the United States, with mortality approaching 50% and a financial burden estimated to exceed $5 billion. Fluid overload, weight gain, and reduced oncotic pressure (low blood proteins) are associated with prolonged need for mechanical ventilation and mortality in patients with ALI/ARDS. Historical studies have provided conflicting evidence for benefits with colloid or diuretic therapy in ALI/ARDS, but recent clinical trials have demonstrated significant improvements in blood oxygen levels. The mechanisms of these benefits are not yet certain, but appear to relate to albumin's (a protein medicine) specific ability to influence injury and inflammation in the lungs, thus improving the ability for the lung to repair and exchange oxygen.

The purpose of this project is to determine the effects of therapies that affect blood proteins on their ability to change the way the lungs and cardiovascular system (heart and blood vessels) function. Special measurements will be taken to understand how these protein medicines change the ability of the lung and whole body to recover from widespread injury, with additional measures of specific heart and lung function. This clinical trial randomizes ALI/ARDS patients with low blood protein levels to receive albumin (a natural blood protein that is known to influence inflammation) or hetastarch (a synthetic blood protein) with diuretic therapy targeted to improve respiratory function. Therapeutic effects on respiratory function and blood oxygen levels, extravascular lung water, oncotic pressure, lung fluid removal, and heart function will be characterized. This trial will advance our understanding of treatment of ALI/ARDS and the factors that affect fluid balance in the lungs of these patients.

Funding Source - FDA Office of Orphan Products Development (OOPD)

ELIGIBILITY:
Inclusion Criteria:

* Consensus clinical definition of ALI or ARDS:

  * Partial pressure of oxygen in arterial blood to the fraction of inspired oxygen (PaO2 / FiO2) ratio ≤ 200 (ARDS) or ≤ 300 (ALI), and;
  * Bilateral infiltrates on chest x-ray, and;
  * No clinical evidence of congestive heart failure, and;
  * Pulmonary artery occlusion pressure (PAOP) ≤ 18 mm Hg, if a pulmonary arterial catheter is present
* Serum total protein concentration < 6.0 g/dL.
* Endotracheal intubation and mechanical ventilation ≥ 24 hours.

Exclusion Criteria:

* Hemodynamic instability within the prior 24 hours: (either of the following)

  * Ongoing fluid resuscitation defined as > 2 liters of crystalloid boluses or > 4 units of blood products transfused in the prior 24-hour period.
  * Vasopressor support exceeding any of the following:
* Dopamine or dobutamine > 5 mcg/kg/min, or in combination at any dose; or
* Any other vasoactive agent (i.e. epinephrine, norepinephrine, phenylephrine)
* Significant renal disease (either of the following at the time of screening):

  * End-stage renal disease, or
  * Renal insufficiency with serum creatinine ≥ 3.0 mg/dL or urine output < 500cc/24 hrs
* Allergy to albumin, hetastarch or furosemide.
* Increased risk for bleeding:

  * Within 72 hours of any surgical procedure requiring use of the operating room, or
  * Any current or previously diagnosed bleeding disorder, or
  * History of any intracranial abnormality (including, but not limited to, intracranial arteriovenous malformations, subdural/subarachnoid/intracerebral hemorrhage, intracranial mass lesions) or traumatic brain injury with Glasgow Coma Scal (GCS) < 9 in the prior 14 days, or
  * Prothrombin time international normalized ratio (INR) > 2.0, partial thromboplastin time (PTT) > 1.5 times control, platelet count < 50,000/cc3
* Risk for worsening pulmonary edema due to systolic heart failure.
* Technical pulse contour analysis limitations:

  * Absence of central venous catheter, clinical arterial vascular disease, severe hypothermia (core temperature < 94°F), weight < 40 kg or > 250 kg, clinically significant bleeding diathesis.
* Failure of the patient or nearest relative to provide informed consent.
* Refusal of the patient's attending physician to provide consent to participate.
* Age < 18 years.
* Pregnancy.
* Inability to quantify urine output (e.g. absence of bladder or bladder catheter).
* Significant hypokalemia (K+ < 3.5 meq/L), hypernatremia (Na+ > 155 meq/L) or hypomagnesemia (Mg < 1.0 meq/L)
* Patient meets criteria for weaning mechanical ventilation:

  * Required FiO2 ≤ 0.40 and positive end-expiratory pressure (PEEP) ≤ 5, and;
  * Spontaneous tidal volumes > 5 ml / kg, and;
  * Spontaneous respiratory rate < 20 / minute, and;
  * Capable of spontaneous ventilation on continuous positive airway pressure (CPAP)=5, pressure support (PS)=5.
* Expected survival ≤ 120 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-01; Primary Completion 2015-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Greg S Martin, MD, MSc, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory Crawford Long Hospital, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Critically ill, mechanically ventilated intensive care patients with Acute Lung Injury (ALI) or Acute Respiratory Distress Syndrome (ARDS) and low blood protein levels were recruited from four hospitals in the Southeast United States between May 1, 2009 and October 31, 2015.
Pre-assignment Details: Not all consented subjects were treated due to changes in eligibility between the consent and treatment periods or subject withdrawal from the study after consent but prior to treatment. 31 individuals gave consent to participate in the study, however, 4 did not begin the study intervention, resulting in 27 who started treatment.
Groups:
- Intravenous 5% Human Albumin: Recipients of continuous infusion intravenous furosemide and administration of intravenous 250 milliliters (mL) 5% human albumin every 8 hours for 5 days
- Intravenous 6% Hetastarch: Recipients of continuous infusion intravenous furosemide and administration of intravenous 250 milliliters (mL) 6% hetastarch every 8 hours for 5 days
Period: Overall Study
Arm/Group | Intravenous 5% Human Albumin | Intravenous 6% Hetastarch
Started | 13 | 14
Completed | 13 | 13
Not Completed | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Intravenous 5% Human Albumin: Recipients of continuous infusion intravenous furosemide and administration of intravenous 250mL 5% human albumin every 8 hours for 5 days
- Intravenous 6% Hetastarch: Recipients of continuous infusion intravenous furosemide and administration of intravenous 250mL 6% hetastarch every 8 hours for 5 days
- Total: Total of all reporting groups
Arm/Group | Intravenous 5% Human Albumin | Intravenous 6% Hetastarch | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (16) | 50 (16) | 49 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 11 | 14 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 9 | 13
  White | 7 | 5 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 13 | 14 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change in Extravascular Lung Water (EVLW)
Description: Quantity of extravascular lung water (EVLW) measured by transpulmonary thermodilution. Higher measurements of EVLW per kilogram of body weight indicate increased lung injury. Normal values for EVLW are thought to be less than 10 mL/kg.
Time Frame: Baseline to Day 5 (120 hours)
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | Intravenous 5% Human Albumin | Intravenous 6% Hetastarch
Number analyzed (Participants) | 13 | 14
mL/kg
  Baseline | 18.5 (7.1) | 17.7 (5.9)
  Hour 120 | 16.0 (7.3) | 15.1 (3.6)

2. Secondary Outcome: Change in Oxygenation (PaO2/FiO2 Ratio)
Description: Change in arterial oxygenation measured by arterial blood gas analysis. The partial pressure of O2 in arterial blood to fraction of inspired oxygen ratio (PaO2/FiO2) is a ratio of partial pressure arterial oxygen to fractional inspired inspired oxygen. This ratio is used as an indicator of hypoxemia (low blood oxygen). A PaO2/FiO2 ratio of 200-300 indicates mild ARDS, 100-200 indicates moderate ARDS, and less than 100 indicates severe ARDS.
Time Frame: Baseline, Day 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Intravenous 5% Human Albumin | Intravenous 6% Hetastarch
Number analyzed (Participants) | 13 | 14
mmHg
  Baseline | 191.3 (53.8) | 157.3 (63.0)
  Day 1 | 213.4 (95.5) | 165.4 (50.8)

3. Secondary Outcome: Ventilator-free Days
Description: The 'ventilator free survival days' in a 30-day period is a previously validated method of comparing groups with respect to mechanical ventilator requirements while adjusting for mortality. This variable represents the number of days in the 30-day period following baseline that the patient is alive and not requiring mechanical ventilation.
Time Frame: Day 30
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Intravenous 5% Human Albumin | Intravenous 6% Hetastarch
Number analyzed (Participants) | 13 | 14
days | 23 [0 to 24] | 23 [0 to 24]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) will be determined daily from enrollment to 72 hours after the last dose of study drug or any study-related procedure. All deaths, unexpected serious adverse events (SAEs), and worsening renal function (as defined as creatinine greater than or equal to 3.0 mg/dL or urine output less than 500cc/24 hrs) will be followed until 30 days after enrollment in this study.
Description: For purposes of this study, an AE is defined as any unfavorable or unintended change in structure, function, signs, or symptoms different from what is expected in the clinical course of an ALI patient and temporally associated with the use of any study drug (albumin, hetastarch or furosemide) or the performance of a study procedure, regardless of any causal relationship to the study.
Arm/Group | Intravenous 5% Human Albumin | Intravenous 6% Hetastarch
All-Cause Mortality (participants affected / at risk) | 1/13 | 3/14
Serious Adverse Events (participants affected / at risk) | 4/13 | 5/14
Other Adverse Events (participants affected / at risk) | 6/13 | 6/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous 5% Human Albumin (N=13) | Intravenous 6% Hetastarch (N=14)
Re-hospitalization (General disorders) | 1 (1) | 0 (0)
Shock (General disorders) | 0 (0) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute hepatic injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bleeding (General disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Focal weakness (General disorders) | 0 (0) | 1 (1)
Acute respiratory distress/failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous 5% Human Albumin (N=13) | Intravenous 6% Hetastarch (N=14)
Systemic hypotension (General disorders) | 4 (7) | 3 (3)
Systemic hypertension (General disorders) | 1 (1) | 0 (0)
Bleeding/coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 4 (6)
Worsening pulmonary edema or lung injury (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Myocardial ischemia (Cardiac disorders) | 0 (0) | 1 (1)
Increase in serum amylase or lipase (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Secondary infection or sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes